CLINICAL TRIAL: NCT00278330
Title: Phase I Trial of Vorinostat (SAHA) in Combination With Alvocidib (Flavopiridol) in Patients With Relapsed, Refractory, or (Selected) Poor Prognosis Acute Leukemia or Refractory Anemia With Excess Blasts-2
Brief Title: Flavopiridol and Vorinostat in Treating Patients With Relapsed or Refractory Acute Leukemia or Chronic Myelogenous Leukemia or Refractory Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00077; MCC 6637; CDR0000656277; R21CA115260 (NIH); U01CA062490 (NIH)
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-04

CONDITIONS: Blastic Phase Chronic Myelogenous Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Relapsing Chronic Myelogenous Leukemia; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — alvocidib; Vorinostat

ARMS (1):
- Arm I (Experimental): Patients will receive a 1-hour infusion of flavopiridol on 5 days in week 1 and vorinostat by mouth three times a day in weeks 1 and 2. Treatment may repeat every 3 weeks for as long as benefit is shown.
  Interventions: Drug: alvocidib; Drug: vorinostat

INTERVENTIONS:
Drug: alvocidib — Given by infusion
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza

SUMMARY:
This phase I trial is studying the side effects and best dose of flavopiridol when given together with vorinostat in treating patients with relapsed or refractory acute leukemia or chronic myelogenous leukemia or refractory anemia. Flavopiridol and vorinostat may cause leukemia cells to look more like normal cells, and to grow and spread more slowly. Vorinostat may also stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving flavopiridol together with vorinostat may be an effective treatment for leukemia or refractory anemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine recommended phase II doses for the combination of flavopiridol and vorinostat in patients with acute leukemia, chronic myelogenous leukemia in blast crisis, or refractory anemia with excess blasts-2.

SECONDARY OBJECTIVES:

I. Determine the safety, toxicity, tolerability, and maximum tolerated dose of this drug regimen.

II. Determine the pharmacodynamic and clinical anti-leukemic effects of this drug regimen.

III. Correlate leukemia gene expression patterns with response in patients treated with this regimen.

OUTLINE: This is an open-label, dose-escalation study of flavopiridol.

Patients receive flavopiridol IV over 1 hour on days 1-5 and oral vorinostat three times daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following:

  * Relapsed or refractory acute leukemia (acute myeloid leukemia [AML], acute lymphoblastic leukemia [ALL], or acute leukemia unclassifiable) following at least one prior systemic treatment
  * Acute leukemia in a patient 60 years or older (no requirement for prior treatment)
  * Acute leukemia that has evolved from a prior myelodysplastic syndrome
  * Chronic myelogenous leukemia (CML) in blast crisis following prior imatinib mesylate therapy
  * Refractory anemia with excess blasts-2 (RAEB-2)
  * No known CNS leukemia
* ECOG performance status 0-2
* WBC < 50,000µL
* Hydroxyurea and/or leukaphereses may be used to lower WBC
* Creatinine =< 1.5 times upper limit of normal (ULN) OR creatinine clearance >= 50 mL/min
* Total bilirubin =< 2 times ULN
* AST/ALT =< 2.5 times ULN
* QTc interval =< 0.470 seconds
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No other condition that would preclude study participation
* At least 3 weeks since prior treatment (expect leukaphereses)
* No valproic acid therapy within the past 2 weeks
* No prior autologous or allogeneic bone marrow or stem cell transplantation
* No hydroxyurea use within the past 24 hours
* No concurrent treatment with other anti-cancer agents or investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
MTD for the combination of alvocidib and vorinostat, assessed by Common Toxicity Criteria version 3.0 | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States